CLINICAL TRIAL: NCT00348062
Title: A Multicenter Evaluation of Methods to Reduce Hyperemia Associated With Bimatoprost Therapy for Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 5177
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost

SUMMARY:
Evaluate the incidence of hyperemia in patients using bimatoprost and to determine if simple interventions reduce its incidence and to assess the value of detailed instruction in increasing patient compliance and willingness to continue bimatoprost therapy, despite the occurrence of hyperemia.

ELIGIBILITY:
Inclusion Criteria:

* · Male or female > 18 years of age

  * No prior use of bimatoprost
  * Diagnosis of open-angle glaucoma or ocular hypertension
  * Ability to provide informed consent and likely to complete all study visits

Exclusion Criteria:

* · Known contraindication to bimatoprost

  * Uncontrolled systemic disease
  * Active ocular disease other than glaucoma or ocular hypertension
  * Required use of ocular medications other than the study medications during the study (intermittent use of artificial tear solutions will be permitted)
  * History of intraocular surgery within the last 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noecker, MD, Principal Investigator — UPMC Eye Center
Locations (1):
- Dr. Noecker, Pittsburgh, Pennsylvania, United States